CLINICAL TRIAL: NCT02332603
Title: Effect of Preoperative Intravenous High Dose Methylprednisolone on Glucose Homeostasis in Patients Scheduled for Total Hip- and Knee-arthroplasty
Brief Title: Effect of Methylprednisolone on Glucose Homeostasis in Patients Undergoing Total Hip- and Knee-arthroplasty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Viktoria Oline Lindberg-Larsen, MD, research assistant, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: HK_VL_08_2014c
Record Dates: First submitted 2015-01-05; First posted 2015-01-07 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Osteoarthrosis
Keywords: Glucocorticoid; Glucose homeostasis; Knee arthroplasty, total; Hip arthroplasty, total
MeSH Terms: conditions — Osteoarthritis | interventions — Methylprednisolone; Methylprednisolone Hemisuccinate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methylprednisolone (Active Comparator): Preoperative single high dose of Solu-Medrol 125 mg iv.
  Interventions: Drug: Methylprednisolone
- Isotonic Sodium Chloride (Placebo Comparator): Preoperative single dose of isotonic Sodium Chloride
  Interventions: Drug: Isotonic Sodium Chloride

INTERVENTIONS:
Drug: Methylprednisolone — Comparison of preoperative single high dose of Methylprednisolone 125 mg iv. and isotonic Sodium Chloride
  Other Names: Solu-Medrol
  Arms: Methylprednisolone
Drug: Isotonic Sodium Chloride — Placebo
  Arms: Isotonic Sodium Chloride

SUMMARY:
This study evaluates the pathophysiological effects of a single dose of Methylprednisolone administered prior to total hip- and knee-arthroplasty surgery. The investigators examine the effect on blood glucose homeostasis.

Half of participants will receive intravenous Solu-Medrol 125 mg, while the other half will receive placebo.

The investigators hypothesize that the glucose homeostasis remains equally stable in the group receiving Methylprednisolone as in the group receiving placebo.

DETAILED DESCRIPTION:
The anti-inflammatory effects of glucocorticoids are well known. The beneficial effects on postoperative pain, postoperative nausea and vomiting are well-documented.

Glucocorticoid might change the glucose metabolism as it induces insulin-resistance. Glucocorticoids are known to reduce the insulin-mediated glucose uptake by reducing the muscle glycogen synthase activity.

The effect of a single high dose of glucocorticoid is poorly described in the literature, and therefore calls for further investigation.

This study is embedded in a primary study registrated as: NCT02319343

For further details please view the EudraCT registration:

EudraCT nr.: 2014-003395-23

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthrosis
* Undergoing total unilateral hip- or knee arthroplasty surgery
* Speak and understand Danish
* Have given informed consent

Exclusion Criteria:

* Revision or bilateral hip- or knee-arthroplasty surgery
* General anaesthesia
* Allergy or intolerance towards Methylprednisolone
* Local or systemic infection
* Permanent systemic treatment with steroids within 30 days preoperatively
* Insulin-dependent diabetes
* Active treatment of ulcer within 3 months preoperatively
* Cancer disease
* Autoimmune disease incl. rheumatoid arthritis
* Pregnant or breast feeding women
* Menopause <1 year

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2015-01; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Changes in plasma blood glucose from baseline (before surgery) to 48 hours after surgery | baseline to 48 hours

SECONDARY OUTCOMES:
Changes in plasma C-peptide from baseline (before surgery) to 48 hours after surgery | baseline to 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Viktoria Lindberg-Larsen, MD, Principal Investigator — Section for Surgical Pathophysiology, Rigshospitalet
Locations (1):
- Bispebjerg Hospital, Copenhagen NV, Denmark

REFERENCES:
- [Background] Husted H. Fast-track hip and knee arthroplasty: clinical and organizational aspects. Acta Orthop Suppl. 2012 Oct;83(346):1-39. doi: 10.3109/17453674.2012.700593. PMID 23205862
- [Background] Kehlet H. Fast-track hip and knee arthroplasty. Lancet. 2013 May 11;381(9878):1600-2. doi: 10.1016/S0140-6736(13)61003-X. No abstract available. PMID 23663938
- [Background] Khan SK, Malviya A, Muller SD, Carluke I, Partington PF, Emmerson KP, Reed MR. Reduced short-term complications and mortality following Enhanced Recovery primary hip and knee arthroplasty: results from 6,000 consecutive procedures. Acta Orthop. 2014 Feb;85(1):26-31. doi: 10.3109/17453674.2013.874925. Epub 2013 Dec 20. PMID 24359028
- [Background] Malviya A, Martin K, Harper I, Muller SD, Emmerson KP, Partington PF, Reed MR. Enhanced recovery program for hip and knee replacement reduces death rate. Acta Orthop. 2011 Oct;82(5):577-81. doi: 10.3109/17453674.2011.618911. Epub 2011 Sep 6. PMID 21895500
- [Background] Abdelmalak BB, Bonilla AM, Yang D, Chowdary HT, Gottlieb A, Lyden SP, Sessler DI. The hyperglycemic response to major noncardiac surgery and the added effect of steroid administration in patients with and without diabetes. Anesth Analg. 2013 May;116(5):1116-1122. doi: 10.1213/ANE.0b013e318288416d. Epub 2013 Apr 4. PMID 23558840
- [Background] Murphy GS, Szokol JW, Avram MJ, Greenberg SB, Shear T, Vender JS, Gray J, Landry E. The effect of single low-dose dexamethasone on blood glucose concentrations in the perioperative period: a randomized, placebo-controlled investigation in gynecologic surgical patients. Anesth Analg. 2014 Jun;118(6):1204-12. doi: 10.1213/ANE.0b013e3182a53981. PMID 24299928
- [Background] de la Motte L, Kehlet H, Vogt K, Nielsen CH, Groenvall JB, Nielsen HB, Andersen A, Schroeder TV, Lonn L. Preoperative methylprednisolone enhances recovery after endovascular aortic repair: a randomized, double-blind, placebo-controlled clinical trial. Ann Surg. 2014 Sep;260(3):540-8; discussion 548-9. doi: 10.1097/SLA.0000000000000895. PMID 25115430
- [Background] Dieleman JM, Nierich AP, Rosseel PM, van der Maaten JM, Hofland J, Diephuis JC, Schepp RM, Boer C, Moons KG, van Herwerden LA, Tijssen JG, Numan SC, Kalkman CJ, van Dijk D; Dexamethasone for Cardiac Surgery (DECS) Study Group. Intraoperative high-dose dexamethasone for cardiac surgery: a randomized controlled trial. JAMA. 2012 Nov 7;308(17):1761-7. doi: 10.1001/jama.2012.14144. PMID 23117776
- [Derived] Lindberg-Larsen V, Kehlet H, Bagger J, Madsbad S. Preoperative High-Dose Methylprednisolone and Glycemic Control Early After Total Hip and Knee Arthroplasty: A Randomized, Double-Blind, Placebo-Controlled Trial. Anesth Analg. 2018 Oct;127(4):906-913. doi: 10.1213/ANE.0000000000003591. PMID 29944516